CLINICAL TRIAL: NCT03586479
Title: Interactive Book Reading to Accelerate Word Learning by Children With SLI
Brief Title: Kindergarten Children Acquiring Words Through Storybook Reading
Acronym: KAWStory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20482; 2R01DC012824 (NIH)
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-06

CONDITIONS: Language Development Disorders
Keywords: Vocabulary
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: Children will be randomly assigned to one of three treatment arms
Who Masked: Outcomes Assessor
Masking Description: Pre- and post-outcome assessments will be performed by an individual blind to arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Testing (Experimental): Children will receive 0 testing (talking) exposures and 6 listening exposures for a total of 6 exposures to each word. This is a listening only condition with minimal testing.
  Interventions: Behavioral: Interactive storybook reading
- Mid Testing (Experimental): Children will receive 2 testing (talking) exposures and 4 listening exposures for a total of 6 exposures to each word. This is a listening and talking condition with mostly listening.
  Interventions: Behavioral: Interactive storybook reading
- High Testing (Experimental): Children will receive 4 testing (talking) exposures and 2 listening exposures for a total of 6 exposures to each word. This is a listening and talking condition with mostly talking.
  Interventions: Behavioral: Interactive storybook reading

INTERVENTIONS:
Behavioral: Interactive storybook reading — Children will be taught 30 words prior to, during, and after reading a commercially available storybook by an adult.
  Other Names: interactive book reading; dialogic reading

SUMMARY:
Children with Specific Language Impairment (SLI) are slower to learn new words than their peers, placing them at risk for academic failure. In this study, we are improving a storybook reading treatment to help Kindergarten children with SLI learn new words. In this study, we compare three versions of book reading that vary in how often children are tested on, meaning asked to talk about, the words they are learning in the book: low vs. mid vs. high testing. We then examine which version of the treatment leads to better learning of the words during treatment and remembering of the words after treatment. We also seek to understand individual differences in treatment outcomes by examining pre-treatment predictors as well as progress during and after treatment.

DETAILED DESCRIPTION:
Children with Specific Language Impairment (SLI) are slower to learn new words than their peers, placing them at risk for academic failure. Our long-term goal is to develop an effective word learning treatment for kindergarten children with SLI, thereby improving their academic and vocational outcomes. During the prior funding period, we successfully taught new words to children with SLI via interactive book reading, a treatment involving an adult reading a storybook to a child and deviating from the text to teach new words. We identified the adequate intensity of the treatment and showed that children with SLI learn an appropriate number of words by the end of 8-weeks of treatment, approximating the number of words learned by typically developing children in prior studies. However, this successful support of short-term word learning revealed new challenges that must be overcome in this renewal to continue to understand and improve long-term word learning by children with SLI. Thus, a second preliminary clinical trial involving 60 kindergarten children with SLI is proposed. Aim 1 addresses the challenge that newly learned words were forgotten once treatment was withdrawn. We attempt to buffer forgetting by comparing different amounts of testing during interactive book reading (low vs. mid vs high testing). Incorporating testing into training is a well-established and highly replicated means of reducing forgetting by adults and typically developing children. Aim 1 will determine whether testing can be harnessed to buffer forgetting by children with SLI under real world conditions. Aims 2 and 3 address the challenge that not all children benefitted equally from interactive book reading. In Aim 2, we identify pre-treatment characteristics of children with SLI that are associated with the slope of learning during treatment or the slope of forgetting post-treatment. Moreover, we select a pre-treatment battery that samples a wide array of skills likely to be associated with learning (language processing, working memory, and episodic memory) or forgetting (overall learning during treatment, decay rate). Aim 2 will provide a foundation for predicting which children will benefit from interactive book reading and will identify which skills are major barriers to long-term word learning by children with SLI. In Aim 3, we classify each child's response at the end of treatment (learner vs. non-learner) and at the end of post-treatment monitoring (rememberer vs. forgetter). Then, we examine earlier performance to determine when treatment and post-treatment outcomes can be predicted. This yields empirically based benchmarks for progress that can be used to tailor the treatment to individual children and establishes the stability of learning and forgetting over time. Overall, this research advances a promising treatment to effectively overcome the significant word learning challenges faced by children with SLI and reveals the contribution of learning and forgetting to language normalization by children with SLI. The results will have impact beyond word learning and SLI because all treatments require boosting learning and buffering forgetting. Thus, the knowledge gained will further catalyze clinical research.

ELIGIBILITY:
Inclusion Criteria:

Eligible for kindergarten enrollment Age 5-6 years Normal hearing Normal nonverbal IQ -- Nonverbal IQ of 85 or higher Language impairment as documented by language score </= 94 on SPELT-3 or </=91 on TNL-2 Vocabulary impairment as documented by a vocabulary score </= 6 on DELV, </= 6 on CELF-4 Word Classes, </= 6 on CCC-2

Exclusion Criteria:

Speaks more than one language Health history indicating neurologic or other disorder that would exclude a diagnosis of SLI (e.g., autism, developmental disability)

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Swinburne Romine, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified pre-treatment test scores and pre-, during, and post-treatment outcome measures will be included as supplemental material to publications. All study information will be shared as supplemental material to publication or upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available as findings are published (in conjunction with publication)
Access Criteria: Data will be open access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Testing | Mid Testing | High Testing
Started | 18 | 14 | 16
Completed | 10 | 11 | 12
Not Completed | 8 | 3 | 4
Not completed — Treatment schedule disrupted during pandemic | 4 | 2 | 2
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Behavioral Issues | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Testing | Mid Testing | High Testing | Total
Number analyzed (Participants) | 10 | 11 | 12 | 33
Age, Continuous [Mean (Standard Deviation); unit: months] — Age is reported in months
  months | 63.4 (5.17) | 63.2 (5.96) | 65.08 (5.37) | 63.97 (5.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 | 13
  Male | 7 | 6 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 10 | 11 | 31
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 9 | 8 | 10 | 27
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 12 | 33
Test of Narrative Language, Second Edition [Mean (Standard Deviation); unit: TNL score] — The Test of Narrative Language-Second Edition "is a comprehensive measure of children's ability to understand and tell stories" (Gillam & Pearson, 2017, page 1). Each child's Narrative Language Ability Index score is reported. To obtain the index, each child's subtest scaled scores are summed and converted to the narrative language ability index . The subtest scaled scores include comprehension and production. The Language Ability Index Score ranges from 50 (less that 1st percentile) to 155 (greater than 99th percentile). Higher values represent a better outcome.
  TNL score | 83.5 (12.01) | 87.55 (12.01) | 88.25 (11.87) | 86.49 (11.60)

OUTCOME MEASURES:

1. Primary Outcome: Change in Definition Scores From Pre- to 12-weeks Post-treatment
Description: This outcome measure indicates the total number of words children responded to correctly at post-test after subtracting the total number of words correct at pre-test. For the definition scores, this includes the total number of words that the child provided correct definitions for at post-test minus the number of words that the child provided correct definition scores at pre-test.
  For each child, there was a total of 30 taught words and 30 untaught words. Thus, for all word learning outcomes the range is 0-30.
  For all assessments of word learning, higher values represent a better outcome. In this study, the subscales are not combined into a total score.
Time Frame: 20 weeks: pre-treatment, treatment (7.5 weeks), 12-weeks post-treatment
Measure: Mean (Standard Deviation); unit: number of words
Arm/Group | Low Testing | Mid Testing | High Testing
Number analyzed (Participants) | 10 | 11 | 12
number of words | 2.50 (2.64) | 3.18 (5.53) | 5.50 (4.10)

2. Secondary Outcome: Change in Naming Scores From Pre- to 12-weeks Post-treatment
Description: This outcome measure indicates the total number of words children responded to correctly at post-test after subtracting the total number of words correct at pre-test. For the naming scores, this included the total number of words that the child provided the correct name for (target word) when given a picture and sentence prompt at post-test, minus the total number of words that the child provided the correct name for at pre-test. For each child, there was a total of 30 taught words and 30 untaught words. Thus, for all word learning outcomes the range is 0-30. For all assessments of word learning, higher values represent a better outcome. In this study, the subscales are not combined into a total score.
Time Frame: 20 weeks: pre-treatment, treatment (7.5 weeks), 12-weeks post-treatment
Measure: Mean (Standard Deviation); unit: number of words
Arm/Group | Low Testing | Mid Testing | High Testing
Number analyzed (Participants) | 10 | 11 | 12
number of words | 6.40 (4.22) | 7.36 (5.52) | 8.50 (6.05)

3. Other Pre Specified Outcome: Change in Untaught Vocabulary
Description: Pre-treatment general vocabulary measures will be re-administered post-treatment. We report the change in number of words defined at pretest and immediate post test. Each child was tested on taught words (words trained during the intervention) and untaught words (words assessed but not trained). Thus, there are four primary outcome scores for word learning: assessments of 1. form and 2. meaning for taught words, and assessments of 3. form and 4. meaning for untaught words.
  For each child, there was a total of 30 taught words and 30 untaught words. Thus, for all word learning outcomes the range is 0-30. For all assessments of word learning, higher values represent a better outcome. In this study, the subscales are not combined into a total score.
Time Frame: 10 weeks: pre-treatment, treatment (7.5 weeks), immediate post-treatment
Population: One child in High Testing Group did not complete immediate post test.
Measure: Mean (Standard Deviation); unit: number of words
Arm/Group | Low Testing | Mid Testing | High Testing
Number analyzed (Participants) | 10 | 11 | 11
number of words | 1.90 (2.42) | 2.64 (2.73) | 0.90 (1.81)

ADVERSE EVENTS:
Time Frame: All participants during the 15 treatment sessions (8 weeks) and during the retention period up to 12 weeks post treatment.
Arm/Group | Low Testing | Mid Testing | High Testing
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/12

LIMITATIONS AND CAVEATS:
We excluded the data from 8 children from analyses whose testing schedules were disrupted due to the 2020 pandemic. These children finished the clinical trial, however, because the primary questions of this study focused on learning rates and forgetting rates, and the schedule for these children differed substantially from the other children, we elected to exclude their data as their treatment schedules would not capture learning and retention rates on the same schedule as other children.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/79/NCT03586479/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT03586479/ICF_002.pdf